CLINICAL TRIAL: NCT07143032
Title: A Comparative Study Between Three Surgical Techniques in Large Angle Exotropia: Bilateral Lateral Rectus Recession With Medial Rectus Resection, Bilateral Medial Rectus Resection and Resection-Transplantation
Brief Title: A Comparative Study Between Three Surgical Techniques in Large Angle Exotropia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Ahmed Abdelraheem, Principle investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-7-4MD
Record Dates: First submitted 2025-08-08; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Exotropia Equal or More Than 50 Prism Diopter
Keywords: exotropia; Recession; Resection; Transplantation
MeSH Terms: conditions — Exotropia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bilateral lateral rectus muscle recession with unilateral medial rectus muscle resection (Active Comparator): patients with large angle exotropia treated by bilateral lateral rectus muscle recession with unilateral medial rectus muscle resection
  Interventions: Procedure: Extropia squint surgery
- bilateral medial rectus muscle resection (Active Comparator): patients with large angle exotropia treated by bilateral medial rectus muscle resection
  Interventions: Procedure: Extropia squint surgery
- unilateral medial rectus muscle resection with lateral rectus muscle transplantation (Active Comparator): patients with large angle exotropia treated by unilateral medial rectus muscle resection with lateral rectus muscle transplantation
  Interventions: Procedure: Extropia squint surgery

INTERVENTIONS:
Procedure: Extropia squint surgery — patients with large angle exotropia will be treated by three different surgical techniques including: 1/ bilateral lateral rectus muscle recession with unilateral medial rectus muscle resection 2/bilateral medial rectus muscle resection, 3/unilateral medial rectus muscle resection with lateral rectus muscle transplantation ,to compare the surgical outcomes between them.

SUMMARY:
This is a randomized comparative interventional study that aims to compare the surgical outcomes of correcting large angle exotropia (≥50 prism diopter) by three different surgical techniques including: 1/ bilateral lateral rectus muscle recession with unilateral medial rectus muscle resection 2/bilateral medial rectus muscle resection, 3/unilateral medial rectus muscle resection with lateral rectus muscle transplantation,

DETAILED DESCRIPTION:
This is a randomized comparative interventional study that will be conducted on patients with large angle exotropia before and after doing surgical correction using three different surgical techniques including : 1/ bilateral lateral rectus muscle recession with unilateral medial rectus muscle resection 2/bilateral medial rectus muscle resection, 3/unilateral medial rectus muscle resection with lateral rectus muscle transplantation ,to compare the surgical outcomes between them.

ELIGIBILITY:
Inclusion Criteria:

* Patients with large-angle exotropia (≥50 prism diopter).

Exclusion Criteria:

1. Patients with an exodeviation angle of less than 50 prism diopter.
2. History of previous strabismus surgery.
3. Restrictive or paretic strabismus or history of botulinum toxin injections for strabismus.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
changes in ocular alignment | at one month, 6 month and one year postoperatively.
  Detect ocular alignment by using Krimsky test to measure angle of deviation in prism diopter

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cifuentes DL, Pineles SL, Demer JL, Velez FG. Surgical success and lateral incomitance following three-muscle surgery for large-angle horizontal strabismus. J AAPOS. 2018 Feb;22(1):17-21. doi: 10.1016/j.jaapos.2017.10.005. Epub 2017 Dec 1. PMID 29199031
- [Background] Talebnejad MR, Johari MK, Khalili MR, Zare M. Supramaximal Recession and Resection Surgery in Large-Angle Strabismus: Outcomes of Large Interventional Case Series Exotropia and Esotropia. J Curr Ophthalmol. 2020 Mar 23;32(1):82-87. doi: 10.4103/JOCO.JOCO_22_20. eCollection 2020 Jan-Mar. PMID 32510018
- [Background] Peters ER, Archer SM. Long-standing, large-angle exotropia in adults. Am Orthopt J. 2007;57:104-6. doi: 10.3368/aoj.57.1.104. PMID 21149163